CLINICAL TRIAL: NCT03114033
Title: TAME Cardiac Arrest Trial: Targeted Therapeutic Mild Hypercapnia After Resuscitated Cardiac Arrest: A Phase III Multi-Centre Randomised Controlled Trial
Brief Title: Targeted Therapeutic Mild Hypercapnia After Resuscitated Cardiac Arrest
Acronym: TAME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Health Research Board, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANZIC-RC/SB001
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Cardiac Arrest; Intensive Care Unit; Therapeutic Mild Hypercapnia; Normocapnia; Mortality; Neurological function
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A Randomised, Parallel Groups, Assessor Blinded, Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted therapeutic mild hypercapnia (Experimental): Target arterial carbon dioxide range of 50-55 mmHg for 24 hours following randomisation
  Interventions: Other: Targeted therapeutic mild hypercapnia
- Targeted normocapnia (Standard care) (Active Comparator): Target arterial carbon dioxide range of 35-45 mmHg for 24 hours following randomisation
  Interventions: Other: Targeted normocapnia (Standard care)

INTERVENTIONS:
Other: Targeted therapeutic mild hypercapnia — Patients allocated to the TTMH protocol will be sedated to achieve moderate to deep sedation (a target Richmond Agitation Scale Score of -4). Arterial blood gases and end- tidal carbon dioxide levels will be measured at baseline and then used to guide respiratory rate adjustments of minute ventilation to remain within the target PaCO2 range of 50-55 mmHg. Arterial blood gases will be repeated every 4 hours for 24 hours following randomisation or if end-tidal carbon dioxide values change >5 mmHg
  Arms: Targeted therapeutic mild hypercapnia
Other: Targeted normocapnia (Standard care) — Patients allocated to the standard care (TN) protocol will be managed according to current practice and in accordance with ILCOR guidelines which recommend maintaining normocapnia in these patients. They will be sedated to achieve moderate to deep sedation (a target Richmond Agitation Scale Score of - 4). Arterial blood gases and end-tidal carbon dioxide levels will be measured at baseline and then used to guide respiratory rate adjustments of minute ventilation to remain within the target PaCO2 range of 35-45 mmHg. Arterial blood gases will be repeated every 4 hours for 24 hours following randomisation or if end-tidal carbon dioxide values change >5 mmHg.
  Arms: Targeted normocapnia (Standard care)

SUMMARY:
The TAME Cardiac Arrest trial will study the ability of higher arterial carbon dioxide (PaCO2) levels to reduce brain damage, comparing giving patients 'normal' to 'slightly higher than normal' blood PaCO2 levels and assessing their ability to return to normal life-tasks. It will be the largest trial ever conducted in heart attack patients in the intensive care unit. This therapy is cost free and, if shown to be effective, will improve thousands of lives, transform clinical practice, and yield major savings.

DETAILED DESCRIPTION:
Cardiac arrest is a common and catastrophic event with substantial human and financial costs. It is well understood that cardiac arrest leads to brain injury. However, what is not widely appreciated is that, after circulation has been restored, cerebral hypoperfusion continues. Ongoing cerebral vasoconstriction and cerebral hypoxia has been demonstrated using technologies that include positron emission tomography, ultrasound, jugular bulb oxygen saturation and cerebral oximetry.

A likely mechanism responsible for sustained early cerebral hypoperfusion relates to impaired cerebrovascular auto-regulation. Such impaired cerebral auto-regulation may make even a normal arterial carbon dioxide tension (PaCO2) (the major physiological regulator of cerebral blood flow) insufficient to achieve and maintain adequate cerebral perfusion and, consequently, cerebral oxygenation. However, PaCO2 is the major determinant of cerebral blood flow and an increased PaCO2 (hypercapnia) markedly increases cerebral blood flow. Moreover, arterial carbon dioxide is modifiable and, as such, is a potential therapeutic target.

The TAME Cardiac Arrest Trial is a definitive phase III multi-centre randomised controlled trial in resuscitated cardiac arrest patients. This trial will determine whether targeted therapeutic mild hypercapnia (TTMH) applied during the first 24 hours of mechanical ventilation in the intensive care unit (ICU) improves neurological outcome at 6 months compared to standard care (targeted normocapnia (TN).

Supported by compelling preliminary data, significant improvements in patient outcomes are achievable with this proposed simple and cost free therapy. Recruiting 1,700 patients, for multiple sites in many countries, this will be the largest trial ever conducted involving resuscitated cardiac arrest patients admitted to the ICU. If the TAME Cardiac Arrest Trial confirms that TTMH is effective, its findings will improve the lives of many, transform clinical practice and yield major economic gains worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years or older)
* Out-of-hospital cardiac arrest of a presumed cardiac or unknown cause
* Sustained ROSC - defined as 20 minutes with signs of circulation without the need for chest compressions
* Unconscious (FOUR-score motor response of <4, not able to obey verbal commands after sustained ROSC) (Appendix D)
* Eligible for intensive care without restrictions or limitations
* Within <180 minutes of ROSC

Exclusion Criteria:

* Unwitnessed cardiac arrest with an initial rhythm of asystole
* Temperature on admission <30oC
* On ECMO prior to ROSC
* Obvious or suspected pregnancy
* Intracranial bleeding
* Severe chronic obstructive pulmonary disorder (COPD) with long-term home oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome | 6 months following enrolment
  Proportion of patients with a favourable (score ≥5) neurological outcome as assessed using the Glasgow Outcomes Score Extended (GOSE) method.

SECONDARY OUTCOMES:
Mortality at intensive care unit discharge | 6 months after randomisation
  Mortality at intensive care unit discharge
Mortality at hospital discharge | 6 months after randomisation
  Mortality at hospital discharge
Health-related Quality of Life (EQ-5D-5L) | 6 months after randomisation
  Health-related Quality of Life (EQ-5D-5L) at 6 months
modified Rankin scale (mRS) | 6 months after randomisation
  modified Rankin scale (mRS) with favourable score of equal to or less than 3
Montreal Cognitive Assessment (MoCA-blind) | 6 months after randomisation
  Montreal Cognitive Assessment (MoCA-blind) at 6 months
Mortality at 6 months | 6 months after randomisation
  Mortality at 6 months
Informant Questionnaire on Cognitive Decline in the Elderly-Cardiac Arrest (IQCODE) | 6 months after randomisation
  IQCODE
Symbol Digit Modality Test | 6 months after randomisation
  SDMT at 6 months

OTHER OUTCOMES:
Quality Adjust Life Years (QALYs) | 6 months after randomisation
  Quality Adjust Life Years (QALYs)
Health economic evaluation | 6 months after randomisation
  Evaluation of hospital and post-discharge estimates of costs at 6 months
Pneumonia | Occurring from enrolment until Day 7 while the participant is in the intensive care unit as reported by treating clinicians.
  Pneumonia as defined by the presence of increased or purulent trachael secretions, new or progressive radiographic infiltrate and a decreased arterial oxygen tension fraction of inspired oxygen ratio of less than 240 mmHg or less than 32 kPa
Sepsis and septic shock | Occurring from enrolment until Day 7 while the participant is in the intensive care unit as reported by treating clinicians.
  Sepsis and septic shock according to the third international consensus definitions for sepsis and septic shock as published in the journal JAMA 2016;315:801-810
Bradycardia | Occurring from enrolment until Day 7 while the participant is in the intensive care unit as reported by treating clinicians.
  Bradycardia requiring pacing
Moderate or severe bleeding | Occurring from enrolment until Day 7 while the participant is in the intensive care unit as reported by treating clinicians.
  Moderate or severe bleeding according to the GUSTO criteria as reported in the journal N Engl J Med 1993;329:673-82
Cooling device-related skin complications | Occurring from enrolment until Day 7 while the participant is in the intensive care unit as reported by treating clinicians.
  Cooling device-related skin complications as defined as being blistering or skin necrosis in areas covered by surface device.
Arrhythmia | Occurring from enrolment until Day 7 while the participant is in the intensive care unit as reported by treating clinicians.
  Arrhythmia that results in haemodynamic compromise (for example ventricular fibrillation and ventricular tachycardia).

CONTACTS AND LOCATIONS:
Overall Officials: Glenn M Eastwood, RN, PhD, Principal Investigator — Monash University
Locations (52):
- Australia (20):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Prince Charles Hospital, Chermside, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Nambour Hospital, Sunshine Coast, Queensland
  - Sunshine Coast University Hospital, Sunshine Coast, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - The Northern Hospital, Epping, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Alfred Health, Melbourne, Victoria
  - Footscray Hospital-Western Health, Melbourne, Victoria
  - Sunshine Hospital-Western Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
- Belgium (3):
  - Cliniques Universitaires de Bruxelles Hospital Erasme, Brussels
  - Ziekenhuis Oost-Limburg AV, Genk
  - University Hospital Ghent, Ghent
- Aarhus University Hospital, Aarhus, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- CHRU Jean Minjoz Besancon, Besançon, Franche Comte, France
- Ireland (4):
  - St. Vincent's University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
- Ospedale San Raffaele, Milan, Italy
- Amsterdam University Medical Centre, Amsterdam, Netherlands
- New Zealand (7):
  - Auckland City Hospital CVICU, Grafton, Auckland
  - Auckland City Hospital DCCM, Grafton, Auckland
  - Middlemore Hospital, Otahuhu, Auckland
  - Christchurch Hospital, Riccarton, Christchurch
  - Wellington Regional Hospital, Newtown, Wellington Region
  - North Shore Hospital, Auckland
  - Rotorua Hospital, Rotorua
- Oslo University Hospital - Ullevål, Oslo, Norway
- King Abdulaziz Medical City, Riyadh, Saudi Arabia
- University Medical Centre Maribor, Maribor, Slovenia
- Sweden (2):
  - Skane Region-Helsingborg, Helsingborg
  - Skane Region Malmö, Malmo
- United Kingdom (8):
  - Queen Alexandra Hospital Portsmouth, Cosham, Portsmouth
  - Royal Victoria Hospital Belfast, Belfast
  - Birmingham University Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Royal Infirmary, Bristol
  - University Hospital Wales, Cardiff
  - Manchester Royal Infirmary, Manchester
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Eastwood GM, Schneider AG, Suzuki S, Peck L, Young H, Tanaka A, Martensson J, Warrillow S, McGuinness S, Parke R, Gilder E, Mccarthy L, Galt P, Taori G, Eliott S, Lamac T, Bailey M, Harley N, Barge D, Hodgson CL, Morganti-Kossmann MC, Pebay A, Conquest A, Archer JS, Bernard S, Stub D, Hart GK, Bellomo R. Targeted therapeutic mild hypercapnia after cardiac arrest: A phase II multi-centre randomised controlled trial (the CCC trial). Resuscitation. 2016 Jul;104:83-90. doi: 10.1016/j.resuscitation.2016.03.023. Epub 2016 Apr 7. PMID 27060535
- [Derived] Melberg MB, Rootwelt SD, Flaa A, Andersen GO, Sunde K, Eastwood G, Olasveengen TM, Qvigstad E. The Effects of Targeted Mild hypercapnia on Right Ventricular Function After Out-of-Hospital Cardiac Arrest: A Substudy of the Targeted Therapeutic Mild Hypercapnia After Resuscitated Cardiac Arrest Trial. Chest. 2025 Nov 24:S0012-3692(25)05796-4. doi: 10.1016/j.chest.2025.11.017. Online ahead of print. PMID 41297587
- [Derived] Melberg MB, Flaa A, Andersen GO, Sunde K, Bellomo R, Eastwood G, Olasveengen TM, Qvigstad E. Effects of mild hypercapnia on myocardial injury after out-of-hospital cardiac arrest. A sub-study of the TAME trial. Resuscitation. 2024 Aug;201:110295. doi: 10.1016/j.resuscitation.2024.110295. Epub 2024 Jun 25. PMID 38936652
- [Derived] Nichol A, Bellomo R, Ady B, Nielsen N, Hodgson C, Parke R, McGuinness S, Skrifvars M, Stub D, Bernard S, Taccone F, Archer J, Neto AS, Trapani T, Ainscough K, Hunt A, Kutsogiannis J, Eastwood GM. Protocol summary and statistical analysis plan for the Targeted Therapeutic Mild Hypercapnia after Resuscitated Cardiac Arrest (TAME) trial. Crit Care Resusc. 2023 Oct 18;23(4):374-385. doi: 10.51893/2021.4.OA2. eCollection 2021 Dec 6. PMID 38046686
- [Derived] Eastwood G, Nichol AD, Hodgson C, Parke RL, McGuinness S, Nielsen N, Bernard S, Skrifvars MB, Stub D, Taccone FS, Archer J, Kutsogiannis D, Dankiewicz J, Lilja G, Cronberg T, Kirkegaard H, Capellier G, Landoni G, Horn J, Olasveengen T, Arabi Y, Chia YW, Markota A, Haenggi M, Wise MP, Grejs AM, Christensen S, Munk-Andersen H, Granfeldt A, Andersen GO, Qvigstad E, Flaa A, Thomas M, Sweet K, Bewley J, Backlund M, Tiainen M, Iten M, Levis A, Peck L, Walsham J, Deane A, Ghosh A, Annoni F, Chen Y, Knight D, Lesona E, Tlayjeh H, Svensek F, McGuigan PJ, Cole J, Pogson D, Hilty MP, During JP, Bailey MJ, Paul E, Ady B, Ainscough K, Hunt A, Monahan S, Trapani T, Fahey C, Bellomo R; TAME Study Investigators. Mild Hypercapnia or Normocapnia after Out-of-Hospital Cardiac Arrest. N Engl J Med. 2023 Jul 6;389(1):45-57. doi: 10.1056/NEJMoa2214552. Epub 2023 Jun 15. PMID 37318140